CLINICAL TRIAL: NCT00223912
Title: Effect of FES- Exercise on Hemostasis in Persons With Chronic Spinal Cord Injury
Brief Title: Effect of Exercise on Blood Coagulation in Persons With Chronic Spinal Cord Injury
Acronym: FES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Kahn, Nighat - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B3168P; 1124-03-0010; MIRB#_00514
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Cardiovascular Disease; Spinal Cord Injury
Keywords: Cardiovascular Disease; Exercise; Functional electrical stimulation; hemostasis; Spinal cord injury
MeSH Terms: conditions — Cardiovascular Diseases; Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Lower-extremity functional electrical stimulation
  Interventions: Device: ERGYS BikeFunctional Electrical Stimulation Ergometry

INTERVENTIONS:
Device: ERGYS BikeFunctional Electrical Stimulation Ergometry — A

SUMMARY:
The purpose of this study is to determine if exercise affects the clotting of blood (hemostasis). The effect of exercise on hemostasis will be determined in persons with spinal cord injury, a population reported to have an increased prevalence of cardiovascular disease (CVD). It is expected that this study will increase our understanding of CVD in persons with SCI, and it will eventually help reduce the occurrence of premature heart disease.

DETAILED DESCRIPTION:
Regular moderate intensity physical exercise decreases platelet aggregability as a consequence of increasing levels of tissue plasminogen activator (tPA) and reducing levels of plasminogen activator inhibitor-1 (PAI-1). In addition, the exercise-associated improvement in the lipid profile and reduction in fat mass may decrease platelet aggregability and blood coagulation, as well as increase fibrinolysis. Thus, it can be hypothesized that physical exercise training has a powerful beneficial impact on blood coagulation and fibrinolysis. Although, regular exercise has been shown to reduce the incidence of CVD and death or causes a regression of symptoms in able-bodied individuals, this salutary effect of prolonged (months) exercise in persons with SCI has not been documented. The present study will evaluate the effects on hemostasis of exercise training in persons with chronic SCI. The effect of exercise on hemostasis will be determined in persons with SCI, a population appreciated to have an increased prevalence of cardiovascular disease (CVD). It is anticipated that this study will ultimately increase our understanding of CVD in this group, and it will eventually help reduce the occurrence of premature macrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

SCI subjects (n=12) with stable chronic, complete paraplegia, (T1 to T10) and quadriplegia (C4 to C8) (for more than 1 year) will be recruited. The paraplegia subjects should be able to transfer independently in/out of a wheelchair.

Exclusion Criteria:

1. Ambulatory persons with SCI
2. Less than 18 years or greater than 65 years old
3. Chronic illness (dialysis)
4. Evidence or history of heart and/or vessel disease (arrhythmias, ischemia at rest)
5. Platelet or coagulation disorders
6. Prescribed use of on aspirin or non-steroidal anti inflammatory drugs
7. Active illness (sepsis, pressure sores)
8. Uncontrolled spasticity
9. Contractures (fixed) in upper extremity/lower extremity Heterotopic ossification at hips, knees, that limit range of motion while seated for FES

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
FES cycle ergometry was performed for 8 sessions. Before and after exercise blood samples were collected and platelet aggregation and blood coagulation analysis were performed. | Before and after exercise (sessions 1 and 8), blood samples were collected.

CONTACTS AND LOCATIONS:
Overall Officials: Nighat Kahn, PhD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- See also: Click here for more information about this study: Effect of FES- Exercise on Hemostasis in Persons with Chronic Spinal Cord Injury — http://www.unitedspinal.org